CLINICAL TRIAL: NCT04590612
Title: The Effects of Mood Symptoms Treatment on Quality of Life and Motor Function in de Novo Parkinson's Disease Patients
Brief Title: Improving Quality of Life in Early Parkinson's Disease
Acronym: PD QOL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Mandar Jog, Principal Investigator, London Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6450
Record Dates: First submitted 2020-09-17; First posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Parkinson Disease; Depression
Keywords: de novo Parkinson disease; depression; quality of life; UPDRS
MeSH Terms: conditions — Parkinson Disease; Depression | interventions — carbidopa, levodopa drug combination; Levodopa; Citalopram

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Carbidopa-Levodopa (Active Comparator): Patients will be randomized to any of the 2 arms. In Levodopa/carbidopa arm, patients will be taking Carbidopa-Levodopa (25-100mg) three times a day for the duration of the study.
  Interventions: Drug: Carbidopa-Levodopa 25 Mg-100 Mg Oral Tablet
- Citalopram (Experimental): Patients will be randomized to any of the 2 arms. In Citalopram arm, patients will be taking Citalopram (20mg) daily for the duration of the study.
  Interventions: Drug: Citalopram

INTERVENTIONS:
Drug: Carbidopa-Levodopa 25 Mg-100 Mg Oral Tablet — 25mg-100mg tablets to be taken orally three times a day on an empty stomach
  Other Names: L-DOPA; l-3,4-dihydroxyphenylalanine; Sinemet
  Arms: Carbidopa-Levodopa
Drug: Citalopram — 20 mg tablet to be taken orally once and at the same time of the day, daily.
  Other Names: Celexa
  Arms: Citalopram

SUMMARY:
The study will examine 30 patients between ages 50-80, newly diagnosed with early-stage Parkinson's Disease. Patients will be randomized to receive either Citalopram or Carbidopa-levodopa. The investigators' primary outcome measure will be change in quality of life over a prospective period of 6 months. Secondary outcome measures will include change in mood state and motor symptoms, as well as comparison of improvement between two treatments.

Primary investigators would also like to collect quantitative electroencephalogram (qEEG) recordings, which is a reading of brain activity as an additional interest of this study. Primary investigators will assess the qEEG recordings for electrophysiological findings before and after interventions.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 50-80 years of age presenting with diagnoses of early stage Parkinson's Disease (UPDRS part III score <20) without a previous treatment trial of either antidepressants or levodopa and able to provide consent.
* Screened positive with depressive symptoms suggestive of an underlying mild to moderate major depressive episode on the PHQ-9 (scores 10-20).

Exclusion Criteria:

* Currently taking an antidepressant (SSRI, SNRI, TCA, MAOi), antipsychotic, or dopaminergic Parkinson medication, or in the last 8 months.
* Tremor with a UPDRS-part III score of 3 or more.
* Currently participating in another clinical trial, which might directly influence findings of this study.
* Inability to provide informed consent.
* Dementia as defined by Montreal Cognitive Assessment (MoCA) score of <24 and/or clinical evidence of dementia.
* A lifetime diagnosis of another mental disorder including bipolar I or II disorder, schizophrenia, schizoaffective disorder, schizophreniform disorder, delusional disorder, moderate and severe alcohol use disorder as per chart review or patient self-report.
* High risk of suicide (e.g. active suicidal ideation and/or current/recent intent or plan) as per self-report or relevant item on the PHQ-9.
* Non-correctable clinically significant sensory impairment.
* Unstable medical illnesses including delirium, uncontrolled diabetes mellitus, hypertension, and hyperlipidemia or cerebrovascular or cardiovascular risk factors that are not under medical management, including QTc>480 on Electrocardiogram.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Difference between two arms in change of Short Form-36 (SF-36) scores | 6 months
  Using a 6-month Randomized Controlled Trial (RCT) intervention study, assess whether Citalopram can improve Quality Of Life (QOL) significantly more than carbidopa-levodopa in early stage Parkinson's disease. This will be measured as a change in SF-36 scores, where the lower scores are associated with more disability. Scores range from 0-100.

SECONDARY OUTCOMES:
Change in Unified Parkinson's Disease Rating Scale (UPDRS) part III motor examination within Citalopram group | 6 months
  Using a 6-months RCT intervention study, assess whether citalopram can improve motor function in early stage Parkinson's disease. Unified Parkinson's Disease Rating Scale part III motor examination indicates higher scores to be associated with more disability. Score ranges from 0 to 132.
Difference between two arms in change of Unified Parkinson's Desease Rating Scale (UPDRS) part III motor examination | 6 months
  Using a 6-months RCT intervention study, assess whether citalopram can improve motor function equally or significantly more than carbidopa-levodopa in early stage Parkinson's disease.Unified Parkinson's Disease Rating Scale part III motor examination indicates higher scores to be associated with more disability. Score ranges from 0 to 132
Difference between two arms in change of Patient Health Questionnaire -9 (PHQ-9) score | 6 months
  Using a 6-months RCT intervention study, assess whether citalopram can improve mood symptoms equally or significantly more than carbidopa-levodopa in early stage Parkinson's disease. Patient Health Questionnaire -9 (PHQ-9) higher score is associated with more disability. Scores range from 0-27.

OTHER OUTCOMES:
quantitative Electroencephalography (qEEG) | at baseline and at 6 months
  Network fragmentation will be analyzed by 5 mins of resting quantitative Electroencephalography (EEG), pre (baseline) and post (6-month followup) treatment. All frequency bands will be analyzed.